CLINICAL TRIAL: NCT00471549
Title: Simvastatin Reduces Plasma Osteoprotegerin in Type 2 Diabetic Patients With Microalbuminuria
Brief Title: Simvastatin Reduces Circulating Osteoprotegerin Levels in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1991/2128
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Dyslipidaemia; Atherosclerosis; Osteoprotegerin; Adhesion molecules; Simvastatin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Dyslipidemias; Atherosclerosis | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Statin (simvastatin)

SUMMARY:
Diabetes is associated with dyslipidaemia leading to generalized atherosclerosis, cardiovascular disease (CVD) and nephropathy. Osteoprotegerin (OPG), a glycoprotein involved in bone homeostasis, has been implicated in the pathogenesis leading up vessel calcification. Furthermore, CVD in diabetics is associated with increased levels of OPG.

Aim: To investigate whether low dose simvastatin treatment (10-20 mg/day) reduces circulating levels of OPG as well as adhesion molecules (VCAM-1; vascular cell adhesion molecule-1, ICAM; intercellular cell adhesion molecule).

DETAILED DESCRIPTION:
Type 2 diabetes is associated with an increased risk of macro- and microvascular complications, resulting from a generalized injury to the vascular endothelium. The pathophysiological mechanisms leading to cardio vascular disease (CVD) in diabetics are not well defined. However, there is accumulating evidence, that damage to vascular smooth muscle cells and endothelial cells partly occur through vessel shear stress, changes in nitric oxide, and increased cytokine levels (i.e. TNF-α: tumour necrosis factor-α and IL-1: interleukin-1). This ultimately results in sclerosis of the basal membrane caused by endothelial cell proliferation and increased vascular permeability, allowing protein to leak into the extra cellular matrix. Atherosclerotic lesions may also arise as a result of accumulation of monocytes and macrophages containing oxidised LDL (foam cells) in the arterial wall. This process is initiated by the expression of adhesion molecules (e.g. VCAM-1; vascular cell adhesion molecule-1, ICAM; intercellular cell adhesion molecule) on the luminal surface of vascular endothelial cells, allowing cellular attachment and migration into the vascular wall.

Osteoprotegerin (OPG), a secreted basic glycoprotein and member of the TNF receptor superfamily, is a soluble receptor activator of nuclear factor-κB (RANK) ligand (RANKL), and TNF-related apoptosis inducing ligand (TRAIL), though with much lower affinity to TRAIL compared to RANKL. OPG works as a decoy-receptor preventing the RANK-RANKL interaction, thereby reducing the biological effect. The RANK-RANKL system induces osteoclast differentiation and activation whereby bone absorption is promoted. Due to its properties as a decoy receptor, OPG antagonizes this effect and inhibits bone loss. In addition to the effects on osteoclasts, the RANK-RANKL system has been proposed to have cardiovascular effects. Thus, activation of the RANK-RANKL system induces VCAM-1 synthesis, prolongs endothelial cell survival, promotes angiogenesis, and reduces TNF-α levels. In contrast, elevated levels of OPG are associated with the severity of CVD, although it is presently unclear whether this association reflects a cause-effect relationship or is purely coincidental.

Cholesterol-lowering therapy with statins reduces cardiovascular mortality and morbidity risk in diabetics and non-diabetic subjects. According to recent studies, statins may have additional, pleiotropic effects and may in fact stabilize atherosclerotic plaques. Experimental data obtained in animal models indicate dose-dependent angiogenetic effects and promotion of vascular structure formation. It is therefore of interest that recent, in vitro studies by Ben-Tahl et al. and Rasmussen et al. suggest that statins may suppress OPG and adhesion molecule production in humans. Thus, umbilical vein endothelial cells and smooth vascular muscle cells incubated with simvastatin and stimulated with TNF-α and IL-1 secreted less OPG than control cells. Under normal circumstances, exposure to cytokines (TNF-α and IL-1) is a powerful stimulus to OPG production in vascular cells and these results therefore seem to support the concept, that simvastatin may ameliorate some of the deleterious effects of inflammation.

This study was conducted to examine the effect of simvastatin treatment on circulating OPG and adhesion molecule levels in a group of type 2 diabetic patients at increased risk for cardiovascular disease (CVD) due to persistent microalbuminuria. Since both OPG and adhesion molecules are associated with CVD and potentially modifiable by statin treatment this could help improve our understanding of potentially pleiotropic effects of statins in reducing CVD.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Persistent microalbuminuria
* Fasting plasma cholesterol > 5.5 mmol/liter
* Fasting plasma triglycerides < 4.5 mmol/liter
* Fasting HbA1c < 10 %
* Fasting serum C-peptide > 0.49 nmol/liter
* Blood pressure < 155/95

Exclusion Criteria:

* Signs of primary kidney disease
* Signs of primary hepatic disease
* Signs of insufficiently treated cardiac disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1991-06; Study Completion 1993-12 (Actual)

PRIMARY OUTCOMES:
Relative reduction in circulating osteoprotegerin levels | 18 weeks

SECONDARY OUTCOMES:
Relative reduction in adhesion molecules (ICAM and VCAM) | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carl E Mogensen, MD, Principal Investigator — Aarhus University Hospital, Department M; Soren Nielsen, MD, PhD, Principal Investigator — Aarhus University Hospital, Department M

REFERENCES:
- [Derived] Nellemann B, Gormsen LC, Dollerup J, Schmitz O, Mogensen CE, Rasmussen LM, Nielsen S. Simvastatin reduces plasma osteoprotegerin in type 2 diabetic patients with microalbuminuria. Diabetes Care. 2007 Dec;30(12):3122-4. doi: 10.2337/dc07-0919. Epub 2007 Sep 5. No abstract available. PMID 17804683